CLINICAL TRIAL: NCT04537442
Title: Clinical Study to Evaluate the Safety and Efficacy of IM21 CAR-T Cells in the Treatment of Elderly Patients With Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Immunochina
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM21 CAR-T cells (Experimental): IM21 CAR-T cells administrated in a dosage to be selected by physician from a specific range.
  Interventions: Drug: IM21 CAR-T cells

INTERVENTIONS:
Drug: IM21 CAR-T cells — IM21 CAR-T cells
  Drug: Fludarabine
  Two days before cell infusion, all patients will be treated with fludarabine for 3 days
  Drug: Cyclophosphamide
  Two days before cell infusion, all patients will be treated with Cyclophosphamide for 3 days
  Other Names:
  Fludarabine Cyclophosphamide

SUMMARY:
This is a single center study to assess the efficacy and safety of IM21 CAR-T cells in adult with R/R multiple myeloma in China.

DETAILED DESCRIPTION:
In this study, about 10 patients with relapsed or refractory multiple myeloma aged ≥60 years were recruited for IM21 CAR-T cell single transfusion therapy. The safety and tolerability of the treatment were evaluated, and the curative effect was initially observed. The research plan includes five stages: screening stage, cell collection stage, chemotherapy pretreatment stage, infusion stage and follow-up stage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory multiple myeloma who had received at least second line regular treatment failure;
2. Age ≥60 years old;
3. The expected survival time is more than 3 months;
4. ECOG score is 0-2;
5. Those who voluntarily participate in the study and sign the informed consent;
6. Hemoglobin (Hb)≥80g/L; Absolute count of neutrophils (ANC) >1×10^9/L Total platelet count (PLT)≥35×10^9/L;
7. left ventricular ejection fraction > 45%.

Exclusion Criteria:

1. High-risk viscera-involved patients: the tumor invaded the gastrointestinal tract, lung, pericardium and one of the great vessels;
2. Those who have graft versus host disease and need to use immunosuppressive agents;
3. Use of systemic steroids in combination within 5 days prior to the blood collection period (except for recent or current use of inhaled steroids);
4. Active hepatitis B or C virus, HIV or other untreated active infected persons;
5. Any circumstance that, in the opinion of the investigator, may increase the risk to the subject or interfere with test results;
6. Patients who use chemotherapy or radiotherapy within 3 days before the blood collection stage.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-09-03 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events within 1 month after CAR-T cell infusion | 30days
  The primary endpoint wasIncidence of adverse events within 1 month after CAR-T cell infusion

SECONDARY OUTCOMES:
Objective Response Rate(ORR) at 90 days | 90days

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, MD, PhD, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang T, Yang Y, Ma L, Feng R, Li J, Zhang C, Bai J, Ding Y, Liu G, Wu F, Lu X, Feng S, Li Z, He T, Li J, Liu H. BCMA-BBZ-OX40 CAR-T Therapy Using an Instant Manufacturing Platform in Multiple Myeloma. J Immunother Cancer. 2024 Sep 23;12(9):e009476. doi: 10.1136/jitc-2024-009476. PMID 39313307
- [Derived] Wang T, He T, Ma L, Yang Y, Feng R, Ding Y, Shan Y, Bu B, Qi F, Wu F, Lu XA, Liu H. Clinical Outcomes of BCMA CAR-T Cells in a Multiple Myeloma Patient With Central Nervous System Invasion. Front Oncol. 2022 May 16;12:854448. doi: 10.3389/fonc.2022.854448. eCollection 2022. PMID 35651792